CLINICAL TRIAL: NCT01468337
Title: Pilot Phase I/II Study of the Treatment of Classic Central Serous Chorioretinopathy With Topical Interferon Gamma-1b
Brief Title: Topical Interferon Gamma-1b for Central Serous Chorioretinopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120013; 12-EI-0013
Record Dates: First submitted 2011-11-05; First posted 2011-11-09 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2014-11

CONDITIONS: Retinal Disease; Macular Disease
Keywords: Central Serous Chorioretinopathy; Interferon-Gamma (IFN-Gamma); Jakstat; Retinal Eye Disease; Macular Eye Disease; CSC
MeSH Terms: conditions — Retinal Diseases; Macular Degeneration; Central Serous Chorioretinopathy | interventions — interferon gamma-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interferon gamma-1b (Experimental): Interferon gamma-1b (Actimmune®, InterMune, Inc, Brisbane, CA 94005) was supplied to participants in single-use dropperettes. A single dropperette contains 1 mL of topical interferon gamma-1b (Actimmune®) at a concentration of 200 µg/mL, which is equivalent to 28 drops. Each drop provides a dose of 7 µg of investigational product.
  All participants will receive interferon gamma-1b for two weeks. Doses of interferon gamma-1b eye drops will be escalated among participants during this initial 2-week period; however, additional doses will be dispensed to participants if needed at Week 4 or after the initial 8-week study period. Participants eligible for additional doses after 8 weeks will be administered the maximum dose of 4 drops 4 times daily for a total daily dose of 112 μg.
  Interventions: Drug: Interferon gamma-1b

INTERVENTIONS:
Drug: Interferon gamma-1b — Participant 1: 2 drops of topical interferon gamma-1b three times daily in the study eye for a daily dose of 42 μg
  Participant 2: 3 drops 3 times daily in the study eye for a daily dose of 63 μg, if the 1st participant's dose is deemed well-tolerated by the investigator at Weeks 1, 2 and 4.
  Participant 3: 3 drops 4 times daily in the study eye for a daily dose of 84 μg, if the 2nd tolerates the daily dose of 63 μg at Weeks 1, 2 and 4.
  Participants 4 and 5: 4 drops 4 times daily in the study eye for a daily dose of 112 μg, if the 3rd tolerates the daily dose of 84 μg at Weeks 1, 2 and 4.
  If the 63, 84 or 112 μg doses are not well-tolerated, subsequent participants will be enrolled at the prior dose level (42, 63 or 84 μg). Well-tolerated is defined as no corneal irritation (e.g., punctuate epithelial keratitis), no coexisting conjunctival erythema and edema, and no signs of more serious toxicities (e.g., intraocular inflammation or lens changes).
  Other Names: Actimmune®

SUMMARY:
Background:

- In the eye disease central serous chorioretinopathy (CSC), fluid collects under the retina at the back of the eye. CSC can resolve on its own, but in some people it lasts for several months or can come back. The fluid buildup during CSC can cause vision loss. The drug interferon gamma-1b can help reduce fluid accumulation in the retina. Researchers want to see if interferon gamma-1b can help treat and prevent vision loss from CSC.

Objectives:

- To see if interferon gamma-1b eye drops are a safe and effective treatment for CSC.

Eligibility:

- Individuals at least 18 years of age who have CSC in at least one eye.

Design:

* Participants will be screened with a physical exam and medical history. They will also have an eye exam and blood tests.
* This study will require at least ten visits to the National Institutes of Health eye clinic over a total of 52 weeks (one year). Most visits will last up to 4 hours.
* Participants will return to the eye clinic 2 days after the first visit and 1, 2, 4, 8, 12, 24, 36 and 48 weeks after starting the study eye drops. These visits will involve blood tests and eye exams.
* Participants will receive the study eye drops at the initial visit. The drops must be used three or four times a day for 2 weeks. They must be stored in a cool place (like a refrigerator). The doses will follow an escalation schedule with the first participant receiving 2 drops three times a day and the last participant receiving 4 drops four times a day. To maximize safety, the most-recently enrolled participant will complete Week 4 before the next participant can enroll (e.g., the second enrolled participant will not be enrolled until the first has completed the Week 4 visit).
* If the CSC does not improve after the first 2 weeks, participants will receive another 2 weeks of eye drops. This set of drops will start 4 weeks after the initial study visit.
* If the CSC does not improve after the 8-week study period, participants may receive additional eye drops at the maximum dose of 4 drops four times daily.
* The study will end for each participant at one year (48 weeks after the initial study visit).

DETAILED DESCRIPTION:
Objective: Central serous chorioretinopathy (CSC) is a retinal disorder characterized by an accumulation of serous fluid under the retina thought to be due to excessive choroidal hyperpermeability. The retinal pigment epithelium (RPE) plays a critical role in removing fluid from the subretinal space. This RPE "pump" is believed to be a key player in the reabsorption of subretinal fluid and maintenance of retinal attachment. Fluid transport assays have examined whether interferon gamma induces changes in fluid transport across human fetal RPE monolayers and showed an increase in fluid absorption from the retinal to the choroidal side of the tissue. An in vivo rodent model of retinal detachment has been used to measure the effect of interferon gamma on re-absorption following retinal detachment and showed that the addition of interferon gamma to the anterior eye surface caused a significant, rapid decrease in retinal detachment volume in the first hour of observation. This pilot study will investigate the safety, tolerability and potential efficacy of serial ocular instillations of topical interferon gamma-1b for classic CSC.

Study Population: Five participants with subretinal fluid due to classic CSC will initially be enrolled. However, up to an additional two participants may be enrolled in order to obtain the five participants to be included in the analysis if any participants withdraw from the study.

Design: In this Phase I/II, non-randomized, prospective, uncontrolled, dose-escalation, single-center pilot study, a series of ocular instillations of topical interferon gamma-1b will be administered in the study eye over a two-week period. If the fluid re-accumulates or increases, participants will be eligible for re-challenging with topical interferon gamma-1b in the study eye at Week 4. Participants will be followed for one year. Participants may be eligible for additional re-challenges after the initial eight week study period ends if their fluid re-accumulates or increases further.

Outcome Measures: The primary outcome measure related to the safety and tolerability of serial ocular instillations of topical interferon gamma-1b will be assessed by the number and severity of adverse events (AEs) related to the investigational product and the number of withdrawals. Secondary efficacy outcomes include changes in best-corrected visual acuity (BCVA), central retinal thickness and maximum lesion volume as measured on optical coherence tomography (OCT), leakage as observed on fluorescein angiograms (FA), autofluorescence patterns as observed on fundus autofluorescence (FAF) imaging and mean macular sensitivity as assessed by microperimetry.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participant must be 18 years of age or older.
* Participant must understand and sign the protocol s informed consent document.
* Female participant of childbearing potential (see Appendix 1 for definition) must not be pregnant or breast-feeding, must have a negative pregnancy test at screening and must be willing to undergo pregnancy tests at scheduled study visits.
* Female participant must be post-menopausal (see Appendix 1), must have had a hysterectomy, have a partner with a vasectomy, be completely abstinent from intercourse or must agree to practice two reliable methods of contraception throughout the course of the study and for six weeks after administration of investigational product. Acceptable methods of contraception include:

  * hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring);
  * intrauterine device;
  * barrier methods (diaphragm, condom) with spermicide; or
  * surgical sterilization (tubal ligation).

EXCLUSION CRITERIA:

* Participant is actively receiving an investigational medication in another research trial that may have unknown effects on CSC as determined by the investigator.
* Participant has evidence of ocular disease other than CSC in the study eye that may confound the outcome of the study (e.g., neovascular age-related macular degeneration).
* Participant has evidence of choroidal neovascularization (CNV) in the study eye.
* Participant is expected to need ocular surgery in the study eye during the eight weeks of the study.
* Participant is expected to need focal laser treatment or photodynamic therapy (PDT) in the study eye during the eight weeks of the study.
* Participant is on medications that enhance RPE pumping of fluid (e.g., acetazolamide).
* Participant is on steroid medication (oral (e.g., prednisone), topical (e.g., hydrocortisone cream) or inhaled (e.g., fluticasone inhaler)).
* Participant has a systemic condition that, in the opinion of the investigator, would preclude participation in the study (e.g., Hypertension not controlled with medications or active infection requiring treatment).
* Participant is allergic to fluorescein dye.
* Participant has multiple sclerosis (MS), as interferon gamma may cause MS exacerbations.
* Participant is on anti-cortisol or anti-androgen medications (e.g., finasteride or mifepristone), as there is some data suggesting that these medications may reduce CSC fluid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Imamura Y, Fujiwara T, Margolis R, Spaide RF. Enhanced depth imaging optical coherence tomography of the choroid in central serous chorioretinopathy. Retina. 2009 Nov-Dec;29(10):1469-73. doi: 10.1097/IAE.0b013e3181be0a83. PMID 19898183
- [Background] Iida T, Kishi S, Hagimura N, Shimizu K. Persistent and bilateral choroidal vascular abnormalities in central serous chorioretinopathy. Retina. 1999;19(6):508-12. doi: 10.1097/00006982-199911000-00005. PMID 10606450
- [Background] Prunte C, Flammer J. Choroidal capillary and venous congestion in central serous chorioretinopathy. Am J Ophthalmol. 1996 Jan;121(1):26-34. doi: 10.1016/s0002-9394(14)70531-8. PMID 8554078

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interferon Gamma-1b
Started | 5
Week 2 | 5
Received Interferon Gamma-1b at Week 4 | 2 (One participant received additional Interferon gamma-1b dosing at Week 4 and after Week 8)
Received Interferon Gamma-1b After Wk 8 | 4 (Two participants had 2 Interferon gamma-1b dosing cycles after Wk 8)
Week 48 | 3 (Two participants did not have a Week 48 visit but completed the study.)
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Severe Ocular Adverse Events Related to the Investigational Product
Time Frame: Week 48
Measure: Number; unit: Adverse Events
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
Adverse Events | 0

2. Primary Outcome: Total Number of Ocular Adverse Events Related to Investigational Product
Time Frame: Week 48
Measure: Number; unit: Adverse Events
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
Adverse Events | 7

3. Primary Outcome: Total Number of Severe Non-ocular Adverse Events Related to the Investigational Product
Time Frame: Week 48
Measure: Number; unit: Adverse Events
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
Adverse Events | 0

4. Primary Outcome: Total Number of Non-ocular Adverse Events Related to the Investigational Product
Time Frame: Week 48
Measure: Number; unit: Adverse Events
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
Adverse Events | 0

5. Primary Outcome: Number of Participants Who Withdrew From the Study
Time Frame: Week 48
Measure: Number; unit: participants
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
participants | 0

6. Secondary Outcome: Changes in Best-corrected Visual Acuity (BCVA) in the Study Eye at Week 2 Compared to Baseline
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
  A positive change value indicates improvement of the outcome. A negative change value indicates worsening of the outcome.
Time Frame: Baseline and Week 2
Measure: Mean (Full Range); unit: ETDRS letters
Units Other Than Participants: Eyes
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
ETDRS letters | 0.4 [-3.00 to 5.00]

7. Secondary Outcome: Changes in Best-corrected Visual Acuity (BCVA) in the Fellow Eye at Week 2 Compared to Baseline
Description: as for outcome 6
Time Frame: Baseline and Week 2
Measure: Mean (Full Range); unit: ETDRS letters
Units Other Than Participants: Eyes
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
ETDRS letters | 0.80 [-2.00 to 7.00]

8. Secondary Outcome: Changes in Best-corrected Visual Acuity (BCVA) in the Study Eye at Week 48 Compared to Baseline
Description: as for outcome 6
Time Frame: Baseline and Week 48
Measure: Mean (Full Range); unit: ETDRS letters
Units Other Than Participants: Eyes
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
ETDRS letters | 2.67 [-3.00 to 13.00]

9. Secondary Outcome: Changes in Best-corrected Visual Acuity (BCVA) in the Fellow Eye at Week 48 Compared to Baseline
Description: as for outcome 6
Time Frame: Baseline and Week 48
Measure: Mean (Full Range); unit: ETDRS letters
Units Other Than Participants: Eyes
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 3
Number analyzed (Eyes) | 3
ETDRS letters | 4.67 [1.00 to 9.00]

10. Secondary Outcome: Changes in the Maximum Subretinal Fluid Volume as Measured on Optical Coherence Tomography (OCT) at Week 2 Compared to Baseline
Time Frame: Baseline and Week 2
Population: Due to lack of effect in other outcome measures, at investigator's discretion, data for this outcome measure was neither collected nor analyzed. As such, zero participants have data for this outcome.
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 0

11. Secondary Outcome: Changes in Central Retinal Thickness as Measured on Optical Coherence Tomography (OCT) at Week 2 Compared to Baseline
Time Frame: Baseline and Week 2
Population: as for outcome 10
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 0

12. Secondary Outcome: Changes in Leakage as Observed on Fluorescein Angiography (FA) at Week 2 Compared to Baseline
Time Frame: Baseline and Week 2
Population: as for outcome 10
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 0

13. Secondary Outcome: Changes in the Autofluorescence Patterns as Observed on Fundus Autofluorescence (FAF) Imaging at Week 2 Compared to Baseline
Time Frame: Baseline and Week 2
Population: as for outcome 10
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 0

14. Secondary Outcome: Changes in Mean Macular Sensitivity as Assessed by Microperimetry at Week 2 Compared to Baseline
Time Frame: Baseline and Week 2
Population: as for outcome 10
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 0

15. Secondary Outcome: Changes in the Maximum Subretinal Fluid Volume as Measured on Optical Coherence Tomography (OCT) at Week 48 Compared to Baseline
Time Frame: Baseline and Week 48
Population: as for outcome 10
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 0

16. Secondary Outcome: Changes in Central Retinal Thickness as Measured on Optical Coherence Tomography (OCT) at Week 48 Compared to Baseline
Time Frame: Baseline and Week 48
Population: as for outcome 10
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 0

17. Secondary Outcome: Changes in Leakage as Observed on Fluorescein Angiography (FA) at Week 48 Compared to Baseline
Time Frame: Baseline and Week 48
Population: as for outcome 10
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 0

18. Secondary Outcome: Changes in the Autofluorescence Patterns as Observed on Fundus Autofluorescence (FAF) Imaging at Week 48 Compared to Baseline
Time Frame: Baseline and Week 48
Population: as for outcome 10
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 0

19. Secondary Outcome: Changes in Mean Macular Sensitivity as Assessed by Microperimetry at Week 48 Compared to Baseline
Time Frame: Baseline and Week 48
Population: as for outcome 10
Arm/Group | Interferon Gamma-1b
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Interferon Gamma-1b
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Gamma-1b (N=5)
Asthenopia (Eye disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 3 (5)
Eye pruritis (Eye disorders) | 2 (2)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 2 (2)
Ocular hypertension (Eye disorders) | 1 (2)
Periorbital oedema (Eye disorders) | 1 (1)
Prostate infection (Infections and infestations) | 1 (1)
Pruritis generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
After study completion, a participant presented with a cataract on 4/12/13 (last study dose:10/3/12 and TOTAL study dosage received: 2758 µg). Although age (58) was consistent with the possibility of cataract, relatedness to drug cannot be ruled out.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes